CLINICAL TRIAL: NCT03192592
Title: Safety and Effectiveness Evaluation of a New Moisturizer Formulation With Antioxidant, Anti-inflammatory and Anti-microbial Effects in the Prevention of a Diabetic Skin Dryness and Complications
Brief Title: Safety and Effectiveness Evaluation of the Apotech® Diabetic Body Moisturizer
Acronym: Apotech
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ANS Pharma (Industry)
Collaborators: Allergisa Pesquisa Dermato-Cosmetica LTDA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 060935_01
Record Dates: First submitted 2017-06-13; First posted 2017-06-20 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Skin Diseases, Metabolic; Skin Care
MeSH Terms: conditions — Skin Diseases, Metabolic

STUDY DESIGN:
Intervention Model Description: This study aim to verify the improvement of texture, elasticity and general appearance of the skin through the application of the cosmetic product Apotech®.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Body moisturizer Apotech® (Experimental): Instructions for use: Massage the product in the body twice a day (morning and evening) with gentle movements until completely absorption. Daily use for 28 days.
  Interventions: Other: Body moisturizer

INTERVENTIONS:
Other: Body moisturizer — Daily body moisturizer application for skin protection and barrier.
  Other Names: Apotech® SkinCare

SUMMARY:
Safety and effectiveness evaluation of a new moisturizer formulation with antioxidant, anti-inflammatory and anti-microbial effects in the prevention of diabetics dry skin and complications.

DETAILED DESCRIPTION:
Safety and effectiveness evaluation of a new moisturizer formulation with antioxidant, anti-inflammatory and anti-microbial effects in the prevention of diabetics dry skin and complications. This study aim to address the target population, subjects with controlled diabetes, to verify the improvement of texture, elasticity, and general appearance of the skin through the application of the cosmetic product Apotech®.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with controlled diabetes
* Any phototype and all skin types

Exclusion Criteria:

* Pregnant women
* Subjects that not match the inclusion criteria

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-06-26 (Actual); Study Completion 2017-07-28 (Estimated)

PRIMARY OUTCOMES:
Skin general appearance | 28 days
  Standard guide for sensory claim substantiation - ASTM
Skin texture | 28 days
  Standard guide for sensory claim substantiation - ASTM
Skin hydration | 28 days
  Standard guide for sensory claim substantiation - ASTM
Skin elasticity and visible cracking | 28 days
  Standard guide for sensory claim substantiation - ASTM

SECONDARY OUTCOMES:
Sensory evaluation of the product | 28 days
  Standard questions

CONTACTS AND LOCATIONS:
Overall Officials: Lucas O. Guerra, MSc, Principal Investigator — Allergisa Pesquisa Dermato-Cosmetica LTDA
Locations (1):
- Allergisa Pesquisa Dermato-Cosmetica, Campinas, São Paulo - Brazil, Brazil

IPD SHARING:
Plan to Share IPD: Undecided